CLINICAL TRIAL: NCT01135693
Title: A Qualitative Study of Service Users' Perspective of Reasons for Detention Under Section 136 of the Mental Health Act 1983 Using Grounded Theory
Brief Title: Service Users' Perspective of Reasons for Detention Under Section 136 of the Mental Health Act 1983
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: South West Yorkshire Partnership NHS Foundation Trust (Other Government)
Responsible Party: Dr Adrian Berry, Interim Care Group Director, South West Yorkshire Partnership NHS Foundation Trust
Other Study IDs: SWYTNHS
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Reasons for Detention Under Mental Health Act 1983
Keywords: Section 136; Mental Health Act 1983; Police; Detention; Failure of community care

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Section 136 of the Mental Health Act (MHA) 1983 allows the police to detain someone in a public place if there are reasons to believe that they may be suffering from a mental disorder and to be in need of care or control. For a significant number of psychiatric patients, detention under section 136 and accessing psychiatric services via the police remains an important, and sometimes the only pathway to care. Approximately 17400 people were detained under section 136 of the MHA 1983 during the year 2005-2006 (Independent Police Complaints Commission, 2008).

Despite the large number of patients accessing mental health services via the police, there is no research available to identify the service users' perspective of what led them to come into contact with police and to identify the reasons for care not being accessed by conventional routes. Royal College Psychiatrists (RCP, 2008) and Independent Police Complaints Commission (IPCC, 2008) found that there was lack of research into the service users' perspective and recommended research into this area.

The investigators have devised this research project to help themselves and the wider research and clinical community understand the service users' perspective of how they came to be detained by the police, whether the community services had failed and explore their views to understand what can be done to improve the service provisions.

Fieldhead hospital, Wakefield provides acute inpatient care for psychiatric patients. Those who are detained under section 136 of the MHA in Wakefield area are taken to a place of safety and following assessment they may be admitted formally or informally to Fieldhead hospital for assessment and treatment. Those who are detained under section 136 of MHA and subsequently admitted as inpatients to Fieldhead hospital will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been detained under Section 136 of the Mental Health Act 1983 and subsequently admitted to Fieldhead Hospital, Wakefield
* Those service users aged between 18 and 65 years
* Those service users who have the capacity to consent to the interview

Exclusion Criteria:

* Those service users who are under 18 years old and over 65 years old at the time of the study
* Service users who are assessed to be incapacitated to consent to the study
* Adults with dementia
* Those who cannot understand and/or speak English sufficiently to participate in interview
* Service user's who are currently experiencing crisis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients who are detained under Section 136 of the Mental Health Act 1983 in Wakefield district and subsequently admitted as inpatients to psychiatric wards at Fieldhead Hospital, Wakefield.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Santhana K Gunasekaran, MBBS MRCPsych LLM, Principal Investigator — South West Yorkshire Partnership NHS Foundation Trust; John H Kent, MBBS FRCPsych, Study Chair — South West Yorkshire Partnership NHS Foundation Trust
Locations (1):
- Fieldhead Hospital, Wakefield, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Kent J, Gunasekaran S. Mentally disordered detainees in the police station: the role of the psychiatrist. Advances in Psychiatric Treatment (2010) 16: 115-123. Docking M, Grace K, Bucke T. Police Custody as a "Place of Safety". Examining the Use of Section 136 of the Mental Health Act 1983. Independent Police Complaints Commission, London (2008). Royal College of Psychiatrists. Standards on the Use of Section 136 of the Mental Health Act 1983 (Council Report CR149). Royal College of Psychiatrists, United Kingdom (2008).
- See also: Sponsoring Organisation — http://www.southwestyorkshire.nhs.uk/
- See also: Directly related study published by principal investigator — http://apt.rcpsych.org/cgi/content/abstract/16/2/115